CLINICAL TRIAL: NCT02819570
Title: Comparison of Two Antibiotic Prophylactic Protocols in Preterm Premature Rupture of the Membranes. A Randomized Prospective, Open Trial
Brief Title: Comparison of Two Antibiotic Prophylactic Protocols in Preterm Premature Rupture of the Membranes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, MD, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0149-15-NHR
Record Dates: First submitted 2016-06-02; First posted 2016-06-30 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Premature Rupture of Membrane
Keywords: early-onset neonatal sepsis; Prophylactic antibiotics; Pregnancy; PPROM; EOS
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Neonatal Sepsis; Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cefuroxime (Experimental): I.V cefuroxime 750 mg*3/d for 2days followed by P.O cefuroxime 500 mgx2/d in addition to P.O roxithromycin 150 mg*2/d for 7 days
  Interventions: Drug: I.V cefuroxime 750 mg*3/d for 2 days; Drug: P.O cefuroxime 500 mgx2/d for 5 days; Drug: P.O roxithromycin 150 mg*2/d for 7 days
- ampicillin (Active Comparator): I.V ampicillin 2 gram x4/d for 2 days followed by P.O moxypen 500 mgx3/d for 5 days in addition to P.O roxithromycin 150 mg*2/d for 7 days
  Interventions: Drug: I.V ampicillin 2 gram x4/d for 2 days; Drug: P.O roxithromycin 150 mg*2/d for 7 days; Drug: P.O moxypen 500 mgx3/d for 5 days

INTERVENTIONS:
Drug: I.V cefuroxime 750 mg*3/d for 2 days
  Arms: cefuroxime
Drug: I.V ampicillin 2 gram x4/d for 2 days
  Arms: ampicillin
Drug: P.O cefuroxime 500 mgx2/d for 5 days
  Arms: cefuroxime
Drug: P.O roxithromycin 150 mg*2/d for 7 days
Drug: P.O moxypen 500 mgx3/d for 5 days
  Arms: ampicillin

SUMMARY:
The objective of the study is to compare a new antibiotic protocol with the current prophylactic treatment in routine use and to evaluate obstetric and neonatal outcome: preterm labor, chorioamnionitis and early onset sepsis

DETAILED DESCRIPTION:
Preterm premature rupture of membranes (PPROM) occurs in approximately 3% of all pregnancies and is associated with approximately one-third of preterm births. The incidence of chorioamnionitis in women with premature rupture of membranes (PROM) at < 27, 28 to 36, and > 37weeks' gestation is 41, 15, and 2%, respectively. Intra-amniotic infection is usually polymicrobial, comprised vaginal or enteric flora including aerobic and anaerobic bacteria and atypical agents, such as Mycoplasma. Group B streptococcus (GBS) has been a frequent pathogen. The American College of Obstetricians and Gynecologists approach to PPROM consists of recommending induction of labor in all women > 34 weeks' gestation. In the absence of intrauterine infection, placental abruption or non-reassuring fetal heart rate, management of women with PPROM < 34 weeks consists of hospitalization from the time of diagnosis until delivery, administration of antenatal corticosteroids, and a 7-day course of antibiotic prophylactic therapy to prolong the latency period. Antibiotic therapy has been associated with significant reductions in chorioamnionitis, deliveries within 48 hours, and early-onset (within 3 days of delivery) neonatal sepsis (EOS). The antibiotic regimen in PPROM usually consists of ampicillin intravenously for 48 hours, followed by oral amoxicillin for 5 days (specifically targeting GBS), and a macrolide targeting atypical agents.

An increase in EOS due to gram negative Enterobacteriaceae have been reported lately with a relative decrease in GBS related EOS . These data may have an impact on the antibiotic regimen used for PPROM. The Local pathogens distribution in cases of EOS and their antibiotic sensitivity profiles in Northern Israel have been explored in a multicenter study There were 27 neonates diagnosed with EOS with positive blood cultures. Aerobic Enterobacteriaceae accounted for 14 cases (52%) and group B streptococcus for 7 cases (26%). Of the Escherichia coli and Klebsiella sp.,only 38% were sensitive to ampicillin. As a result the most effective antibiotic protocol to cover those pathogens is required. The purpose of the current study is to compare a new antibiotic protocol with the current prophylactic treatment in use and to evaluate pregnancy and neonatal outcome.

The diagnosis of preterm premature rupture of membranes (PPROM) is clinical, and is based on visualization of amniotic fluid in the vagina of a woman who presents with a history of leaking fluid. Laboratory tests as "Amniosure" can be used to confirm the clinical diagnosis when it is uncertain.

Women who meet the study criteria and have signed inform consent will be randomly divided in two groups to receive prophylactic antibiotic treatment as follow:

1. I.V ampicillin 2 gram x4/d for 2 days followed by P.O moxypen 500 mgx3/d for additional 5 days+ P.O roxithromycin 150 mg*2/d for 7 days
2. I.V cefuroxime 750 mg*3/d for 2days followed by P.O cefuroxime 500 mgx2/d + P.O roxithromycin 150 mg*2/d for 7 days

A course of corticosteroids will be given to all women participating in the study

Expectant management:

1. Vital signs *3/day
2. Uterine tenderness evaluation
3. Complete Blood Count + C-reactive protein every second day
4. Urine culture and GBS recto-vaginal swab
5. Fetal heart monitoring*6 /d
6. Sonography evaluation every 2-3 days
7. Vaginal swab once a week
8. Fetal movements follow up

Labor induction will be conducted at 34 weeks of gestation If chorioamnionitis is suspected amniocentesis should be considered or expeditious delivery

ELIGIBILITY:
Inclusion Criteria:

* Women with PPROM between 24+0 and 34+0 weeks of gestation who are suitable for conservative management

Exclusion Criteria:

* P-PROM>34 weeks of gestation
* Suspected fetal distress or chorioamnionitis
* Active labor
* Drug allergy to one of the study regiments
* Immune deficiency
* Multiple pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
EARLY NEONATAL SEPSIS - positive blood culture | within 3 days of delivery
  Number of Participants with early neonatal sepsis
latency period | from date of randomization until the date of delivery assessed up to 10 weeks
  time in days
Chorioamnionitis rate | from day of randomization until date of clinical/laboratory chorioamnionitis diagnosis assessed up to 10 weeks
  rate of positive cultures

SECONDARY OUTCOMES:
Neonatal weight | at delivery
  grams
Apgar score | 1 minute 5 minute
  score from 0 to 10

OTHER OUTCOMES:
Number of participants with adverse events as assessed by umbilical cord acid-based analysis<7 | at delivery
  cord ph analysis at delivery (units of moles per liter)
Neonatal intensive care unit (NICU) admission duration | days since delivery until rerelease from NICU, assessed up to 6 month
  days from admission until rerelease from NICU assessed up to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Maya Wolf, MD, Principal Investigator — 1Department of Obstetrics & Gynecology, Galilee Medical Center, 2Faculty of Medicine in the Galilee, Bar Ilan University, Nahariya, Israel
Locations (1):
- Galil Medical Center, Nahariya, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mercer BM. Preterm premature rupture of the membranes: current approaches to evaluation and management. Obstet Gynecol Clin North Am. 2005 Sep;32(3):411-28. doi: 10.1016/j.ogc.2005.03.003. PMID 16125041
- [Background] Newton ER. Chorioamnionitis and intraamniotic infection. Clin Obstet Gynecol. 1993 Dec;36(4):795-808. doi: 10.1097/00003081-199312000-00004. PMID 8293582
- [Background] Sperling RS, Newton E, Gibbs RS. Intraamniotic infection in low-birth-weight infants. J Infect Dis. 1988 Jan;157(1):113-7. doi: 10.1093/infdis/157.1.113. PMID 3335795
- [Background] Practice bulletins No. 139: premature rupture of membranes. Obstet Gynecol. 2013 Oct;122(4):918-930. doi: 10.1097/01.AOG.0000435415.21944.8f. PMID 24084566
- [Background] Carlan SJ, O'Brien WF, Parsons MT, Lense JJ. Preterm premature rupture of membranes: a randomized study of home versus hospital management. Obstet Gynecol. 1993 Jan;81(1):61-4. PMID 8416463
- [Background] Turnbull DA, Wilkinson C, Gerard K, Shanahan M, Ryan P, Griffith EC, Kruzins G, Stamp GE. Clinical, psychosocial, and economic effects of antenatal day care for three medical complications of pregnancy: a randomised controlled trial of 395 women. Lancet. 2004 Apr 3;363(9415):1104-9. doi: 10.1016/S0140-6736(04)15893-5. PMID 15064028
- [Background] Roberts D, Dalziel S. Antenatal corticosteroids for accelerating fetal lung maturation for women at risk of preterm birth. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004454. doi: 10.1002/14651858.CD004454.pub2. PMID 16856047
- [Background] Harding JE, Pang J, Knight DB, Liggins GC. Do antenatal corticosteroids help in the setting of preterm rupture of membranes? Am J Obstet Gynecol. 2001 Jan;184(2):131-9. doi: 10.1067/mob.2001.108331. PMID 11174492
- [Background] Kenyon S, Boulvain M, Neilson JP. Antibiotics for preterm rupture of membranes. Cochrane Database Syst Rev. 2013 Dec 2;2013(12):CD001058. doi: 10.1002/14651858.CD001058.pub3. PMID 24297389
- [Background] Mercer BM, Miodovnik M, Thurnau GR, Goldenberg RL, Das AF, Ramsey RD, Rabello YA, Meis PJ, Moawad AH, Iams JD, Van Dorsten JP, Paul RH, Bottoms SF, Merenstein G, Thom EA, Roberts JM, McNellis D. Antibiotic therapy for reduction of infant morbidity after preterm premature rupture of the membranes. A randomized controlled trial. National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. JAMA. 1997 Sep 24;278(12):989-95. PMID 9307346
- [Background] Workowski KA, Berman S; Centers for Disease Control and Prevention (CDC). Sexually transmitted diseases treatment guidelines, 2010. MMWR Recomm Rep. 2010 Dec 17;59(RR-12):1-110. PMID 21160459
- [Background] Grigsby PL, Novy MJ, Sadowsky DW, Morgan TK, Long M, Acosta E, Duffy LB, Waites KB. Maternal azithromycin therapy for Ureaplasma intraamniotic infection delays preterm delivery and reduces fetal lung injury in a primate model. Am J Obstet Gynecol. 2012 Dec;207(6):475.e1-475.e14. doi: 10.1016/j.ajog.2012.10.871. Epub 2012 Oct 23. PMID 23111115
- [Background] Wolf MF, Miron D, Peleg D, Rechnitzer H, Portnov I, Salim R, Keness Y, Reich D, Ami MB, Peretz A, Koshnir A, Shachar IB. Reconsidering the Current Preterm Premature Rupture of Membranes Antibiotic Prophylactic Protocol. Am J Perinatol. 2015 Nov;32(13):1247-50. doi: 10.1055/s-0035-1552935. Epub 2015 May 29. PMID 26023907
- [Derived] Sgayer I, Francis YN, Miron D, Shprits E, Sheffer VF, Rechnitzer H, Lowenstein L, Wolf MF. Compared perinatal outcomes of two prophylactic antibiotic regimens for preterm premature rupture of membranes: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 May;5(5):100900. doi: 10.1016/j.ajogmf.2023.100900. Epub 2023 Feb 13. PMID 36791845
- [Derived] Wolf MF, Sgayer I, Miron D, Krencel A, Sheffer VF, Idriss SS, Sammour RN, Peleg D, Shachar IB, Rechnitzer H, Bornstein J. A novel extended prophylactic antibiotic regimen in preterm pre-labor rupture of membranes: A randomized trial. Int J Infect Dis. 2020 Jul;96:254-259. doi: 10.1016/j.ijid.2020.05.005. Epub 2020 May 11. PMID 32407901